CLINICAL TRIAL: NCT01386788
Title: European Survey: Risk of Cyanide Poisoning in Smoke Inhalation, Symptoms, Key Treatment and Outcome (RISK)
Brief Title: European Survey: Risk of Cyanide Poisoning in Smoke Inhalation
Acronym: RISK
Status: Completed | Type: Observational
Sponsor: Dr. Ernst MW Koch (Other)
Responsible Party: Sponsor-Investigator, Dr. Ernst MW Koch, Dr, Dr. Ernst MW Koch
Other Study IDs: EML015722-600; 2009-010202-11 (Other: EudraCT No)
Record Dates: First submitted 2011-06-27; First posted 2011-07-01 (Estimated); Results first posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-08

CONDITIONS: Smoke Inhalation Patients
Keywords: Smoke, cyanide, closed space fires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Smoke Inhalation patients: Closed space fire, Soot deposits, Altered mental status Blood specimen before intravenous antidote treatment (cyanide measurement) Known delay between end of smoke exposure and blood sampling
  Interventions: Other: There is no intervention planned (observational)

INTERVENTIONS:
Other: There is no intervention planned (observational) — No intervention foreseen

SUMMARY:
Cyanide poisoning is commonly viewed as a rare but dramatic event, occurring in industrial or laboratory settings as the result of accidental releases of hydrogen cyanide (HCN) gas (e.g. in the case of fire) or salts in the case of suicide attempts.

In fact, cyanide poisoning is considerably more common than is generally appreciated. Multiple clinical and post-mortal studies have demonstrated that HCN contributes to the toxicity of fire smoke.

Cyanide acts primarily through its strong affinity for the iron-containing heme moiety, binding to numerous critical enzyme systems in the body and rendering them inactive. Of late, increasing attention has been paid to the relationship of cyanide and nitric oxide. The interactions appear to be complex, with cyanide inducing nitric oxide production by binding to N-methyl-D-aspartate (NMDA) receptors, as well as binding to nitric oxide synthase. The latter may be overcome by the presence of nitric oxide synthase inhibitors.

Probably, the majority of the cyanide poisoning cases are due to smoke inhalation in closed-space fires.

So far, there are no clear data available on the prevalence of cyanide poisoning in smoke inhalation.

This information would be of great interest for all emergency physicians since a proven or supposed cyanide poisoning does not only requires an intensive supportive care, including the administration of supplemental oxygen and artificial ventilation, blood pressure support, and anticonvulsants, but also a rapid administration of a cyanide antidote.

Therefore, it is the goal of this survey to assess the prevalence of cyanide poisoning in smoke inhalation victims. Only the data of patients with a cyanide measurement before specific antidote treatment will be included

DETAILED DESCRIPTION:
Cyanide poisoning is commonly viewed as a rare but dramatic event, occurring in industrial or laboratory settings as the result of accidental releases of hydrogen cyanide (HCN) gas (e.g. in the case of fire) or salts in the case of suicide attempts.

In fact, cyanide poisoning is considerably more common than is generally appreciated. Multiple clinical [1-4] and post-mortal studies [5-10] have demonstrated that HCN contributes to the toxicity of fire smoke.

Cyanide acts primarily through its strong affinity for the iron-containing heme moiety, binding to numerous critical enzyme systems in the body and rendering them inactive [11]. Of late, increasing attention has been paid to the relationship of cyanide and nitric oxide. The interactions appear to be complex, with cyanide inducing nitric oxide production by binding to N-methyl-D-aspartate (NMDA) receptors [12], as well as binding to nitric oxide synthase. The latter may be overcome by the presence of nitric oxide synthase inhibitors.

Probably, the majority of the cyanide poisoning cases are due to smoke inhalation in closed-space fires.

So far, there are no clear data available on the prevalence of cyanide poisoning in smoke inhalation.

This information would be of great interest for all emergency physicians since a proven or supposed cyanide poisoning does not only requires an intensive supportive care, including the administration of supplemental oxygen and artificial ventilation, blood pressure support, and anticonvulsants, but also a rapid administration of a cyanide antidote.

Therefore, it is the goal of this survey to assess the prevalence of cyanide poisoning in smoke inhalation victims. Only the data of patients with a cyanide measurement before specific antidote treatment will be included.

ELIGIBILITY:
Inclusion Criteria:

* Closed space fire, Soot deposits, Altered mental status
* Blood specimen before intravenous antidote treatment (cyanide measurement)
* Known delay between end of smoke exposure and blood sampling
* Malaise and/or Headache and/or Altered mental status in fire workers

Exclusion Criteria:

* Pregnancy
* Multiple trauma, Blast
* Patient pronounced dead at scene without resuscitation attempt
* Patient in whom the time elapsed between the end of exposure and blood sampling is greater than 2 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with smoke inhalation
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zilker, Prof., Study Chair — TU München; Carlo A Locatelli, Prof, Study Chair — IRCCS Fondazione Maugeri; Frédéric Baud, Prof, Study Chair — Hôpital Lariboisière; Guillermo Burillo-Putze, Prof, Study Chair — Universidad de Teneriffe; Jean-Philippe Fauville, Dr, Study Chair — To be added; Francois Levy, Dr, Study Chair — To be added
Locations (2):
- Germany (2):
  - Prof. Dr. Götz Geldner, Ludwigsburg
  - Prof. Th. Zilker, München

REFERENCES:
- [Result] Geldner G, Koch EM, Gottwald-Hostalek U, Baud F, Burillo G, Fauville JP, Levi F, Locatelli C, Zilker T. Report on a study of fires with smoke gas development : determination of blood cyanide levels, clinical signs and laboratory values in victims. Anaesthesist. 2013 Aug;62(8):609-16. doi: 10.1007/s00101-013-2209-3. Epub 2013 Aug 7. PMID 23917894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 102 patients were enrolled, data of 100 patients were evaluated
Groups:
- Smoke Inhalation Victims: Smoke inhalation victims included civil victims and fire workers as specified in the inclusion criteria were observed.
Period: Overall Study
Arm/Group | Smoke Inhalation Victims
Started | 102
Completed | 100
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Smoke Inhalation Victims
Number analyzed (Participants) | 102
Age, Continuous [Mean (Full Range); unit: years] | 49.4 (19) [20 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 63

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival After 24 Hours
Description: Number of participants who survived at 24 hours after smoke inhalation were reported.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Smoke Inhalation Victims
Number analyzed (Participants) | 102
participants | 96

2. Primary Outcome: Serum Cyanide Levels
Time Frame: blood sampling within 2 hours after smoke inhalation
Population: All recruited patients that met all inclusion criteria including blood sampling for cyanide serum level
Measure: Number; unit: participants
Arm/Group | Smoke Inhalation Victims
Number analyzed (Participants) | 100
participants
  <1.1 mcmol/l | 25
  1.2 - 5 mcmol/l | 49
  >5 - 10 mcmol/l | 5
  >10- 20 mcmol/l | 7
  >20- 40 mcmol/l | 4
  >40- 100 mcmol/l | 7
  >100 mcmol/l | 3

ADVERSE EVENTS:
Description: Serious and other [non-serious] adverse events were not collected/assessed.
Groups:
- Smoke Inhalation Victim: Smoke inhalation victims included civil victims and fire workers as specified in the inclusion criteria were observed
Arm/Group | Smoke Inhalation Victim
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
General limitations of observational study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No